CLINICAL TRIAL: NCT04932304
Title: Kognitiv Trening Etter Hjerneslag: Effekter og Mekanismer #2015/1282
Brief Title: Cognitive Training After Stroke : Effects and Mechanisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Lars Tjelta Westlye, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015/1282
Record Dates: First submitted 2021-06-08; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active stimulation (Active Comparator): Participants recieving active trancranial direct current stimulation (tDCS) Parameters: 20 minutes anodal tDCS 1mA. Two times a week, for three weeks. Anode placed at F3, cathode placed at right cerebellum.
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Sham stimulation (Placebo Comparator): Participants recieving passive / sham trancranial direct current stimulation (tDCS) Two times a week, for three weeks. Anode placed at F3, cathode placed at right cerebellum.
  Interventions: Device: Sham Transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS)
  Arms: Active stimulation
Device: Sham Transcranial direct current stimulation (tDCS) — Sham Transcranial direct current stimulation (tDCS)
  Arms: Sham stimulation

SUMMARY:
Stroke is a major cause of severe cognitive and physical disability. Despite the high and increasing incidence, and large health, economic, social and personal consequences, studies designed to remedy cognitive impairments and improve rehabilitation care following stroke are lacking. A promising line of research have shown that weak electrical current (tDCS) can be a safe, cost-effective, and potent treatment when combined with other rehablitational approaches.

The underlying mechanism is assumed that tDCS facilitates neuronal signaling, improving plasticity and facilitating rehablitational outcome. But further research is needed to better understand the mechanisms at hand, and to better evaluate the potential clinical utility.

The scope for the current project is to investigate both cognitive and neuronal effects of tDCS in combination with cognitive training , with the ultimate goal to improve current rehabilitational healthcare. To achieve this we will use multimodal MRI, EEG, and a comprehensive battery of neuropsychological asessment, to describe and evaluate the effect of tDCS in rehabilitation purposes.

DETAILED DESCRIPTION:
Participants are randomly assigned to either active or sham condition, using codes provided by the manufacturer and implemented by an in-house Matlab script, pseudo-randomizing participants while maintaining balance in groups of 20. tDCS stimulation is applied at six occasions for each participant, with a minimum of 48 hours between stimulations, aiming at an average of two stimulations per week. Stimulation current is1000 μA, stimulation time was 20 min for the active group with a ramp-up time of 120 s and fade-out time of 30 s. The current intensity is limited to 1 mA to limit the risk of adverse events due to the electrical stimulation. The sham stimulation consists of ramp-up followed by 40 s of active stimulation and then fade-out, following factory settings.

Cognitive training will be done by the computerized working memory training program (Cogmed Systems AB, Stockholm, Sweden) consisting of 25 online training sessions. In this study, to increase feasibility, we utilize 17 sessions over a period of three to four weeks, corresponding to approximately five weekly training sessions. On average, we aim at two training sessions combined with tDCS per week with a minimum of one day between each tDCS session. The remaining CCT sessions are performed at home.

Neuropsychological assessments and MRI assessments are conducted three times: at baseline 1, after a waiting period of 2-4 weeks (baseline 2, before intervention) and immediately post intervention. Self-reported symptoms of fatigue and depression are assessed at five time points, before, during and after completing intervention.

ELIGIBILITY:
Inclusion Criteria:

- MR/CT revealing ischemic or hemorrhagic damage (stroke).

Exclusion Criteria:

* History of illness or damage to the CNS, besides stroke.
* <18 years of age
* Extensive cognitive decline or dementia
* Severe psychiatric disorders
* Substance or alcohol abuse
* Contraindications for MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Evidence of change in neural activity in attentional-related brain areas after receiving anodal tDCS, as measured with functional MRI | One and a half year
  Change in activation patterns during multiple object tracking (MOT) at first baseline, before initiating training (second baseline, on average 4 weeks after baseline measure), and after a three-week intervention (post-intervention assessment)
Evidence of structural changes after receiving anodal tDCS, as measured with structural MRI | One and a half year
  Structural MRI
Evidence of increased attentional and working memory capacity after receiving anodal tDCS | One and a half year
  Rate of improvement in Cogmed tasks

SECONDARY OUTCOMES:
Evidence of increased attentional capacity after receiving anodal tDCS | One and a half year
  Performance change in The Theory of Visual Attention (TVA) computerized paradigm.

OTHER OUTCOMES:
Evidence of change in fatigue severity after receiving tDCS | One and a half year
  Fatigue Severity Scale (FSS), a seven-point Likert scale on subjective fatigue severity/impact. 9 items scored from 1 (less symptoms) to 7 (most severe symptoms). Scores are reported as mean scores, lowest possible mean = 1, highest possible mean = 7.
Evidence of change in symptoms of depression after receiving tDCS | One and a half year
  Patient Health Questionnaire (PHQ-9), self-reported depressive symptoms. Scale consists of 9 items, scored from 0 (not at all) to 3 (nearly every day). Scores are reported as sum scores, range 0 (less symptoms) - 27 (more symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Lars T. Westlye, Ph.D, Study Director — University of Oslo
Locations (2):
- Norway (2):
  - Oslo University Hospital Ullevål, Oslo
  - Oslo University Hospital, Oslo